CLINICAL TRIAL: NCT01212237
Title: Phase I Study of Dose Response of Functionally Critical Brain Regions for Brain Radiotherapy
Brief Title: Dose Response of Functionally Critical Brain Regions for Brain Radiotherapy
Status: Withdrawn | Type: Observational
Why Stopped: There were no patients enrolled on this study.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 1003010928
Record Dates: First submitted 2010-06-22; First posted 2010-09-30 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Brain Tumors
Keywords: glioma; meningioma; anaplastic astrocytoma
MeSH Terms: conditions — Brain Neoplasms; Glioma; Meningioma; Astrocytoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- fMRI Evaluation: All patients will undergo the following standard imaging and radiotherapy procedures will be performed for each patient:
  1. Standard MRI for radiotherapy treatment planning which takes about 60 minutes.
  2. Radiotherapy treatment simulation with CT.
  3. Radiotherapy treatment planning
  4. Radiotherapy treatment
  5. Routine follow-up every 3 months after the radiotherapy.
  Special Procedures.
  The following special imaging and radiotherapy procedures will be performed for each patient:
  1. fMRI (30 minutes)
  2. The 3MS examination, administered every 3 months during routine follow-up for one year after the completion of the radiotherapy.
  Interventions: Procedure: fMRI Evaluation

INTERVENTIONS:
Procedure: fMRI Evaluation — Functional magnetic resonance imaging (fMRI) uses MR imaging to measure the tiny metabolic changes that take place in an active part of the brain. fMRIs are used for many reasons, for example, to determine precisely which part of the brain is handling critical functions such as thought, speech, movement and sensation, to help assess the effects of stroke, trauma or degenerative disease (such as Alzheimer's) on brain function, and to guide the planning of surgery and radiation therapy.
  Other Names: fMRI

SUMMARY:
Normal tissue response is critical for brain radiotherapy, especially for dose escalation which carries with it an increased incidence of radiation-induced brain injury. Although radiation toxicity and limiting dose for anatomically critical structures of the brain have been well studied and documented, little is known for functionally critical brain regions and treatment of cognitive sequelae of cranial radiotherapy is limited. The objective of this clinical protocol is to accumulate preliminary data for future studies aiming to quantify dose response for functionally critical brain regions for brain radiotherapy. We plan to achieve this objective by correlating the radiation-induced complications and radiological changes with the radiation dose to the selected functionally critical brain regions for 25 patients. Each participating patient will receive brain fMRI to identify brain regions for processing visual, working memory and language functions. The image co-registration algorithm developed previously by our group will be used to co-register these regions on the CT scans for radiotherapy treatment planning for radiation dose calculation. Radiation-induced changes in cognitive functions will be evaluated using the modified mini mental status exam (3MS) and fMRI during the routine follow-up. The knowledge derived from this study might significantly improve the quality of life and allow safer dose escalation for patients receiving brain radiotherapy.

DETAILED DESCRIPTION:
Research Question:

Our goal is to answer the following three research questions in this study:

1. What is the dose response curve (degree of radiation complications/radiological changes vs. radiation dose) for brain regions involved in the processing of visual, language and working memory functions?
2. What is the limiting dose for these functionally critical brain regions that can be applied to radiotherapy treatment planning to minimize (e.g., less than 5%) the possibility of radiation-induced injury?
3. Can brain fMRI be used to guide the radiotherapy treatment planning to minimize the dose to functionally critical brain regions and evaluate treatment responses of these regions?

Research Method:

Imaging before radiotherapy: For each patient, active stimulation and resting fMRI examinations will be performed in addition to standard anatomic MRI for brain radiotherapy. Activation maps of regions involved in visual, language and working memory functions will be generated from the fMRI scans and the patient's responses on of the working memory task (i.e., the N-Back task) will be recorded during the fMRI studies. The MRI and fMRI will, combined, take approximately 90 minutes - 60 minutes for the standard MRI and 30 minutes for the fMRI. The activation maps will be overlaid onto the FLAIR MRI images, imported into the radiotherapy treatment planning system and co-registered with the simulation CT scan.

Radiotherapy and routine follow-up: Functionally critical areas in the fMRI activation maps will be separately contoured as critical organs but will not be considered for plan optimization. Dose volume histograms (DVHs) of functionally critically brain regions will be calculated and documented. Each patient will receive fractionated brain radiotherapy according to the treatment plan and will be followed up with every three months after radiotherapy.

Follow-up evaluations: The 3MS examination will be administered prior to initiation of treatment onset and every three months after treatment during routine follow-up to screen neuropsychological functions. Anatomic MRI (standard) and brain fMRI (research) will be acquired at 6 months after radiotherapy to determine the radiological and functional changes in regions involved in the processing of visual, language and working memory functions.

Minimizing the interference of tumor recurrence or progression: Two actions will be taken to minimize the interference of tumor recurrence or progression with the evaluation of performance alterations caused by radiation. First, patient inclusion will be restricted to patients with slow growing tumors, e.g., meningioma, low grade glioma and anaplastic astrocytoma so that the chance for tumor recurrence or progression is small. Secondly, patients who develop disease progression at any of the post-radiotherapy follow-ups will be excluded from the study, as it would not be possible to distinguish the effects of disease progression from radiotherapy side effects on the fMRI or the 3MS examination, and the findings would not be interpretable.

Dose Response Analysis: Logistic regression analysis will be used to assess the likelihood of complications to functionally critical brain regions as a function of radiation dose. The dependent variable will be the binary indicator that identifies patients' manifesting complications (decline of 3MS examination score and N-Back test, radiological/functional changes identified on MRI and fMRI) attributed to radiation exposure. The logistic regression model will include relevant subject level factors (e.g., age, gender, baseline Karnofsky performance status, tumor location, recent seizures, anti-epleptic medications) as covariates. The fitted logistic normal tissue complication probability (NTCP) model will permit estimation of the probability of significant complications associated with any radiation dose to the area, allowing the limiting dose to be calculated as the dose expected to induce complication with an acceptable probability (e.g., 5%).

Incorporation of limiting dose for radiotherapy treatment planning: The limiting dose from the above "Dose Response Analysis" will be used for IMRT re-planning considering the functionally critical brain regions. The optimization goal is to minimize the dose to functionally critical brain regions while maintaining similar PTV (planning target volume) coverage and keeping dose to the critical structures within accepted tolerance. DVHs of the functionally critical brain regions, PTV and all other critical structures will be compared for both treatment plans with and without considering the functionally critical brain regions. A Wilcoxon matched pair signed rank test will be performed to compare the plans in terms of calculated NTCP of critical organs. The McNemar test will be used to compare plans with and without dose constraints of functional areas in terms of yield rate (i.e., the proportion of patients for whom the IMRT plan was successfully devised).

The primary study endpoint of this study is normal tissue complication. The primary objective of this study is to determine the dose response curve and limiting dose for functionally critically brain regions for brain radiotherapy. The second objective of this study is to investigate the accuracy of active stimulation or resting state fMRI for avoidance of the functionally critical brain regions for radiotherapy treatment planning of brain tumors and for evaluating the treatment responses of these critical regions.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically confirmed diagnosis of slow growing brain tumors that requires radiotherapy, e.g., meningioma, low grade glioma or anaplastic astrocytomas.

  2. A diagnostic contrast enhanced CT/MRI demonstrating the lesion prior to registration.

  3. Karnofsky performance status ≥60. 4. Ability to undergo MR imaging with the use of Gadolinium contrast. 5. Ability to undergo brain fMRI. 6. Patient must sign a study specific informed consent form. Patients who cannot provide consent due to cognitive impairment will not be enrolled in the study. The investigators will follow the recently published guidelines (Binder & Guze, Am. J. Psy., 155, 1649-1650, 1998) to assess the subject's understanding of the procedure and his/her decision making capacity,.

Exclusion Criteria:

* 1. Any condition including allergy to Gadolinium contrast, metallic implants or cardiac pace makers that makes the candidate ineligible for MR imaging. These criteria will be determined by an MRI research screening form signed by the subject.

  2. Any condition including taking anti-anxiety medicines such as Benzodiazepines or requiring sedative to overcome claustrophobia that makes the candidate ineligible brain fMRI.

  3. Karnofsky performance status of ≤60 4. Prior history of radiation therapy to the brain 5. Pregnancy 6. Significant medical or neurological disorders that would affect the outcome of the evaluations and/or make a successful MRI/fMRI unduly difficult 7. Major psychiatric conditions, whether medicated or unmedicated, as such conditions can affect the validity of the evaluations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with brain tumors (astrocytoma, meningioma, low grad glioma)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-05-14 (Actual); Primary Completion 2013-04-13 (Actual); Study Completion 2013-04-13 (Actual)

PRIMARY OUTCOMES:
fMRI to Measure Functional Changes of Criticial Brain Regions Over Time | pre-radiation therapy and 6 months post radiation therapy
  fMRI screening at baseline and 6 months after the completion of radiation therapy to observe the original functionality of the brain (pre-radiation therapy) and the functionality of the brain after radiation therapy. If the radiation has damaged any functional areas, the difference in performance will be evident in the 6 month fMRI.

SECONDARY OUTCOMES:
MMSE - expanded (Mini-Mental Status Examination)- to Document Changes in Functionality of Critical Brain Regions | pre-radiation therapy, 3, 6, 9, 12 months post-radiation therapy
  The expanded MMSE (mini-mental status exam) routinely used to screen the overall cognitive functions of patients following brain radiotherapy. The MMSE will help to track brain function at a great interval than the fMRI. It will show changes in the brain over time.

CONTACTS AND LOCATIONS:
Overall Officials: Jenghwa Chang, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States